CLINICAL TRIAL: NCT01515943
Title: Effectiveness of Home-Based Therapy for Symptomatic Convergence Insufficiency
Brief Title: Convergence Insufficiency Treatment Study (CITS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CITS; 2U10EY011751 (NIH)
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Convergence Insufficiency
Keywords: Convergence insufficiency
MeSH Terms: conditions — Ocular Motility Disorders | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Computer-based therapy (CBT) (Active Comparator): The CBT group will be assigned active home-based computer vergence/accommodative therapy (15 minutes/day) plus placebo yoked prism flipper therapy (5 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Interventions: Other: Active home-based computer vergence/accommodative therapy; Procedure: Placebo yoked prism flippers
- Near target push-up (NTP) (Active Comparator): The NTP group will be assigned placebo home-based computer vergence/accommodative therapy (5 minutes/day) plus near target push-ups (15 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Interventions: Procedure: Near target push-ups; Other: Placebo home-based computer vergence/accommodative therapy
- Placebo (Placebo Comparator): The placebo group will be assigned placebo home-based computer vergence/accommodative therapy (15 minutes/day) plus placebo yoked prism flipper therapy (5 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Interventions: Other: Placebo home-based computer vergence/accommodative therapy; Procedure: Placebo yoked prism flippers

INTERVENTIONS:
Other: Active home-based computer vergence/accommodative therapy — At enrollment, subjects will be prescribed 15 minutes/day of active home-based computer therapy for 5 days/week during the 12 week treatment phase. Active home-based computer therapy will be provided the Home Therapy System (HTS) computer software and will include both fusional vergence and accommodative therapy. Subjects will perform the computer therapy while wearing red/blue glasses and accommodative therapy will be performed using the HTS accommodative flippers. Please refer to the procedures manual for further details.
  Other Names: Home Therapy System (HTS, Home Vision Therapy, Inc.)
  Arms: Computer-based therapy (CBT)
Procedure: Near target push-ups — At enrollment, subjects will be prescribed 15 minutes/day (3 sessions of 5 minutes each) of near target push-ups (NTP) for 5 days/week during the 12-week treatment phase. An alphabet pencil will be used as the target and an index card placed in the background will provide physiological diplopia control. With the pencil positioned at arm's length directly between the subject's eyes, the subject will slowly bring the pencil toward his/her nose while focusing on the small letter on the pencil. When the subject is no longer able to maintain a single image of the pencil, he/she will slowly move the target away from the nose until the pencil becomes single again. This procedure will be repeated several times. Please refer to the procedures manual for further details.
  Other Names: Pencil push-ups
  Arms: Near target push-up (NTP)
Other: Placebo home-based computer vergence/accommodative therapy — At enrollment, subjects will be prescribed either 5 minutes/day (NTP group) or 15 minutes/day (Placebo group) of placebo home-based computer therapy for 5 days/week during the 12 week treatment phase. Placebo computer-based therapy will be provided by the Home Therapy System (HTS) computer software. The vergence procedures are similar to the active version, however, the tasks will be modified to ensure no demand on the vergence system and no accommodative therapy is included in the placebo version. Please refer to the procedures manual for further details.
  Other Names: Home Therapy System (HTS, Home Vision Therapy, Inc.)
  Arms: Near target push-up (NTP); Placebo
Procedure: Placebo yoked prism flippers — Subjects will be prescribed 5 minutes/day of placebo yoked prism flipper therapy for 5 days/week during the 12 week treatment phase. This procedure utilizes a 4 pd base right/4 pd base left prism flipper and "Accommodative Hopping Cards". Subjects view the text on the card through the prisms at 40 cm, perform the appropriate task and then flip the prism flipper to the other side after each word before proceeding to the next line. Please refer to the procedures manual for further details. The task remains constant, but the nature of the procedure changes with time:
  * Weeks 1-4: View the target through prism flippers
  * Weeks 5-8: Wear red-blue filter glasses while viewing the text through prism flippers
  * Weeks 9-12: Wear polaroid glasses while viewing the text through prism flippers
  Arms: Computer-based therapy (CBT); Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of home-based computer therapy for symptomatic convergence insufficiency (CI) compared to traditional home-based near target push-ups and placebo treatment.

DETAILED DESCRIPTION:
Convergence insufficiency (CI) is a common and distinct binocular vision disorder that affects approximately 4% of school age children and adults in the United States. Convergence insufficiency is often associated with symptoms such as frequent loss of place while reading, loss of concentration, having to re-read, reading slowly, poor comprehension, sleepiness, blurred vision, diplopia, headaches, and/or eyestrain. A recently completed randomized clinical trial, the Convergence Insufficiency Treatment Trial (CITT), demonstrated that a 12-week program of office-based vergence/ accommodative therapy with home reinforcement was more effective than home-based near target pencil push-ups, home-based computer accommodative therapy plus pencil push-ups, or office-based placebo therapy in treating the symptoms and signs associated with symptomatic CI in children 9 to 17 years of age.

While the home-based therapies in the CITT were not as effective as office-based vergence/accommodative therapy there was some improvement noted. Currently, many eye care professionals only offer home-based therapy, while others suggest passive treatment with base-in prism. At a Pediatric Eye Disease Investigator Group (PEDIG) meeting (Tampa, January 2009), the results of a poll of attendees indicated that a large majority of pediatric ophthalmologists continue to recommend home-based near target push-ups as the initial treatment approach for children with symptomatic CI in spite of the CITT results.

There are significant differences in contact time, complexity, and cost between office-based and home-based therapy for CI. Many clinicians believe that the less costly and less complex treatment option should be attempted first. Although home-based therapy using computer software is becoming more popular, no prospective data are available to demonstrate the effectiveness of home-based vision therapy using computer software compared to home-based near target push-ups or home-based placebo computer therapy. A prospective clinical trial is therefore needed to determine the effectiveness of home-based computer therapy for symptomatic CI compared to traditional home-based near target push-ups and placebo treatment.

The current study is a multi-center randomized clinical trial to evaluate the effectiveness of home-based computer vergence/accommodative therapy and home-based near target push-ups in children 9 to <18 years of age with symptomatic CI.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 9 to <18 years
2. Patient has access to a computer with a CD/DVD drive and internet access for the next 12 weeks
3. Best-corrected visual acuity of ≥20/25 in each eye at distance and near
4. Exophoria at near at least 4 pd greater than at distance
5. Reduced positive fusional convergence at near (<20 pd or fails Sheard's criterion that the PFV measures less than twice the magnitude of the near phoria). PFV is recorded as the prism magnitude where vision is first blurred (or break if no blur is reported).
6. Near point of convergence of ≥6 cm break
7. Randot Preschool stereoacuity of at least 400 seconds of arc
8. CI Symptom Survey score ≥16
9. No use of a plus add for near or base-in prism for at least 2 weeks preceding enrollment
10. Patient must be wearing appropriate refractive correction (spectacle or contact lenses) for at least 2 weeks prior to enrollment if refractive error is present (based on a cycloplegic refraction within the last 6 months) that meets the following:

    * Myopia more than -0.75D spherical equivalent (SE) in either eye
    * Hyperopia more than +2.00D SE in either eye
    * SE anisometropia >1.00D
    * Astigmatism > 1.00D or > 1.50D of meridional difference in either eye Refractive correction for patients meeting the above refractive error criteria must meet the following guidelines:
    * SE anisometropia must be within 0.25D of the full anisometropic correction.
    * Astigmatism cylinder must be within 0.50D of full correction and axis must be within 5 degrees.
    * For hyperopia, the spherical component can be reduced by up to 1.50D at investigator discretion provided the reduction is symmetrical and results in residual (i.e., uncorrected) SE hyperopia that does not exceed +2.00D.
    * For myopia, the SE must be within 0.25D of the full myopic correction.
11. Parent and patient understand the protocol and are willing to accept randomization.
12. Parent has home phone (or access to phone) and is willing to be contacted by Jaeb Center staff.
13. Relocation outside of area of an active PEDIG site within the next 15 months is not anticipated.

Exclusion Criteria:

1. ≥2 logMAR line difference in best-corrected visual acuity between the two eyes
2. Constant or intermittent exotropia at distance; constant exotropia at near
3. Any esotropia at distance or near
4. Distance exophoria > 10 pd
5. History of strabismus surgery
6. Anisometropia ≥2.00D in any meridian between the eyes
7. Prior intraocular or refractive surgery
8. Primary vertical heterophoria greater than 1 pd
9. Diseases known to affect accommodation, vergence, and ocular motility such as multiple sclerosis, Graves orbitopathy, myasthenia gravis, diabetes mellitus, or Parkinson disease
10. Current use of any ocular or systemic medication known to affect accommodation or vergence such as anti-anxiety agents (e.g., Librium or Valium), anti-arrhythmic agents (e.g., Cifenline, Cibenzoline), anti- cholinergics (e.g., Motion sickness patch (scopolamine), bladder spasmolytic drugs (e.g., Propiverine), hydroxychloroquine, chloroquine, phenothiazines (e.g., Compazine, Mellaril, Thorazine), tricyclic antidepressants (e.g., Elavil, Nortriptyline, Tofranil)
11. Near point of accommodation >20 cm in the right eye
12. Manifest or latent nystagmus evident clinically
13. History of chronic headaches unrelated to reading activity
14. Active symptomatic allergic conjunctivitis
15. Developmental disability, mental retardation, attention deficit hyperactivity disorder (ADHD), or learning disability diagnosis that in the investigator's discretion would interfere with treatment or evaluation
16. Household member or sibling already enrolled in the CITS OR previously enrolled in the CITT
17. Household member is an eye professional, ophthalmic technician, ophthalmology or optometry resident, orthoptist, or optometry student, or employed in an eye care setting
18. Acquired brain injury
19. Previous office- or home-based vision therapy, orthoptics, home-based near- target push-ups, pencil push-ups, or home-based computer therapy

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell M Scheiman, OD, Study Chair — Jaeb Center for Health Research; Darren L Hoover, MD, Study Chair — Jaeb Center for Health Research
Locations (2):
- United States (2):
  - Everett & Hurite Ophthalmic Association, Cranberry TWP, Pennsylvania
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group. Home-Based Therapy for Symptomatic Convergence Insufficiency in Children: A Randomized Clinical Trial. Optom Vis Sci. 2016 Dec;93(12):1457-1465. doi: 10.1097/OPX.0000000000000975. PMID 27575992
- [Derived] Scheiman M, Kulp MT, Cotter SA, Lawrenson JG, Wang L, Li T. Interventions for convergence insufficiency: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 2;12(12):CD006768. doi: 10.1002/14651858.CD006768.pub3. PMID 33263359

RESULTS

PARTICIPANT FLOW:
Groups:
- Computer-based Therapy (CBT): The CBT group will be assigned active home-based computer vergence/accommodative therapy (15 minutes/day) plus placebo yoked prism flipper therapy (5 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Active home-based computer vergence/accommodative therapy: At enrollment, subjects will be prescribed 15 minutes/day of active home-based computer therapy for 5 days/week during the 12 week treatment phase. Active home-based computer therapy will be provided the Home Therapy System (HTS) computer software and will include both fusional vergence and accommodative therapy. Subjects will perform the computer therapy while wearing red/blue glasses and accommodative therapy will be performed using the HTS accommodative flippers. Please refer to the procedures manual for further details.
  Placebo yoked prism flippers: Subjects will be prescribed 5 minutes/day of placebo yoked prism flipper therapy for 5 days/week during the 12 week treatment
- Near Target Push-up (NTP): The NTP group will be assigned placebo home-based computer vergence/accommodative therapy (5 minutes/day) plus near target push-ups (15 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Near target push-ups: At enrollment, subjects will be prescribed 15 minutes/day (3 sessions of 5 minutes each) of near target push-ups (NTP) for 5 days/week during the 12-week treatment phase. An alphabet pencil will be used as the target and an index card placed in the background will provide physiological diplopia control. With the pencil positioned at arm's length directly between the subject's eyes, the subject will slowly bring the pencil toward his/her nose while focusing on the small letter on the pencil. When the subject is no longer able to maintain a single image of the pencil, he/she will slowly move the target away from the nose until the pencil becomes single again. This procedure will be repeated several times.
- Placebo: The placebo group will be assigned placebo home-based computer vergence/accommodative therapy (15 minutes/day) plus placebo yoked prism flipper therapy (5 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Placebo home-based computer vergence/accommodative therapy: At enrollment, subjects will be prescribed either 5 minutes/day (NTP group) or 15 minutes/day (Placebo group) of placebo home-based computer therapy for 5 days/week during the 12 week treatment phase. Placebo computer-based therapy will be provided by the Home Therapy System (HTS) computer software. The vergence procedures are similar to the active version, however, the tasks will be modified to ensure no demand on the vergence system and no accommodative therapy is included in the placebo version. Please refer to the procedures manual for further details.
  Placebo yoked prism flippers: Subjects will be prescribed 5 minutes/day of placebo yoked prism flipper therapy for 5
Period: Overall Study
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Started | 75 | 85 | 44
Completed | 69 | 69 | 31
Not Completed | 6 | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Near Target Push-up (NTP): The NTP group will be assigned placebo home-based computer vergence/accommodative therapy (5 minutes/day) plus near target push-ups (15 minutes/day) for a total of 20/minutes per day, 5 days per week for the 12-week treatment phase.
  Near target push-ups: At enrollment, subjects will be prescribed 15 minutes/day (3 sessions of 5 minutes each) of near target push-ups (NTP) for 5 days/week during the 12-week treatment phase. An alphabet pencil will be used as the target and an index card placed in the background will provide physiological diplopia control. With the pencil positioned at arm's length directly between the subject's eyes, the subject will slowly bring the pencil toward his/her nose while focusing on the small letter on the pencil. When the subject is no longer able to maintain a single image of the pencil, he/she will slowly move the target away from the nose until the pencil becomes single again. This procedure will be repeated several times. Please refer to the pr
- Total: Total of all reporting groups
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo | Total
Number analyzed (Participants) | 75 | 85 | 44 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 85 | 44 | 204
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (2.4) | 12.6 (2.5) | 12.3 (2.3) | 12.4 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 26 | 118
  Male | 29 | 39 | 18 | 86
Region of Enrollment [Number; unit: participants]
  United States | 75 | 85 | 44 | 204

OUTCOME MEASURES:

1. Primary Outcome: Treatment Group Comparison of the Percentage of Participants Classified as an Overall Success at 12 Weeks - HB-C Versus HB-PU
Description: Pairwise treatment group comparison (HB-C versus HB-PU) of the percentages of participants meeting success criteria using binomial regression adjusting for baseline covariates of CISS score (<28 points vs ≥ 28 points), mean NPC break (<10 cm vs ≥ 10 cm), and mean PFV blur (≥ 15 PD vs <15 PD) using linear contrasts with Bonferroni adjustment for multiple comparisons (Type I error rate = 2.5%).
  Overall success was defined as meeting all of the following criteria at 12 weeks:
  1. Convergence Insufficiency Symptom Survey (CISS): 12-week score <16 points and at least 9-point improvement from baseline at 12 weeks
  2. Near point of convergence (NPC) break: 12-week/baseline mean NPC break <0.763 and a mean 12-week NPC break <6 cm
  3. Positive fusional vergence (PFV) blur: 12-week/baseline mean PFV blur >1.419 and a mean 12-week PFV break >15 pd
Time Frame: 12 weeks after randomization (baseline)
Population: The analysis was limited to participants who completed the 12-week visit within the pre-specified analysis window (10 to 18 weeks, inclusive).
Measure: Count of Participants; unit: Participants
Groups:
- Computer-based Therapy (CBT): Prescribed 15 minutes of active computer vergence/accommodative therapy (CVAT) and 5 minutes of placebo flipper exercises, 5 days per week for 12 weeks to be performed at home.
- Near Target Push-up (NTP): Prescribed 15 minutes (in full or split into three 5-minute intervals) of a well-defined near target push-up (NTP) procedure and 5 minutes of placebo computer vergence/accommodative therapy (CVAT), 5 days per week for 12 weeks to be performed at home.
- Placebo: Prescribed 15 minutes of placebo computer vergence/accommodative therapy (CVAT) and 5 minutes of placebo flipper exercises, 5 days per week for 12 weeks to be performed at home.
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 31
Participants | 16 | 15 | 5
Statistical Analysis 1: Comparison: Computer-based Therapy (CBT) vs Near Target Push-up (NTP); The primary outcome was success at 12 weeks. The sample size was computed to have 90% power to detect a treatment group difference between the HB-C versus HB-PU groups, assuming true population success percentages of 30% and 15% for the HB-C and HB-PU groups, respectively, with a type I error rate of 2.5%. The treatment group comparison was adjusted for baseline covariates of CISS score (<28 points vs ≥28 points), mean NPC break (<10 cm vs ≥10 cm) and mean PFV blur (≥15 pd vs <15 pd); Test type: Superiority or Other; p = 0.56, Biniomial regression — Linear contrasts performed with a type I error rate of 2.5% based on a Bonferroni adjustment (overall type I error rate of 5% for 2 pairwise treatment group comparisons); Adjusted for baseline covariates of CISS score, mean NPC break and mean PFV blur. Linear contrasts performed with Bonferroni adjustment (alpha=0.025); Risk Difference (RD) = -4, 97.5% CI 2-sided [-19 to 11] — Negative values for the treatment group difference favor the HB-PU group. Results of the treatment group comparison are adjusted for baseline covariates of CISS, mean NPC break and mean PFV blur

2. Primary Outcome: Treatment Group Comparison of the Percentage of Participants Classified as an Overall Success at 12 Weeks - HB-C Versus HB-P
Description: Pairwise treatment group comparison (HB-C versus Placebo) of the percentages of participants meeting success criteria using binomial regression adjusting for baseline covariates of CISS score (<28 points vs ≥ 28 points), mean NPC break (<10 cm vs ≥ 10 cm), and mean PFV blur (≥ 15 PD vs <15 PD) using linear contrasts with Bonferroni adjustment for multiple comparisons.
  Overall success was defined as meeting all of the following criteria at 12 weeks:
  1. Convergence Insufficiency Symptom Survey (CISS): 12-week score <16 points and at least 9-point improvement from baseline at 12 weeks
  2. Near point of convergence (NPC) break: 12-week/baseline mean NPC break <0.763 and a mean 12-week NPC break <6 cm
  3. Positive fusional vergence (PFV) blur: 12-week/baseline mean PFV blur >1.419 and a mean 12-week PFV break >15 pd
Time Frame: 12-weeks after randomization (baseline)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 31
Participants | 16 | 15 | 5
Statistical Analysis 1: Comparison: Computer-based Therapy (CBT) vs Placebo; The primary outcome was success at 12 weeks. The sample size was computed to have 90% power to detect a treatment group difference between the HB-C versus HB-P groups, assuming true population success percentages of 30% and 10% for the HB-C and HB-PU groups, respectively, with a type I error rate of 2.5%. The treatment group comparison was adjusted for baseline covariates of CISS score (<28 points vs ≥28 points), mean NPC break (<10 cm vs ≥10 cm) and mean PFV blur (≥15 pd vs <15 pd); Test type: Superiority or Other; p = 0.52, Binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 5, 97.5% CI 2-sided [-12 to 22] — Positive values for the treatment group difference favor the HB-C group. Results of the treatment group comparison are adjusted for baseline covariates of CISS, mean NPC break and mean PFV blur

3. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria Based on CI Signs/Symptoms at 12 Weeks by Treatment Group
Description: The number of subjects classified as a success based on signs/symptoms at the 12-week visit. Success is based on the Convergency Insufficiency Symptom Survey (CISS) defined as improvement of 9 or more points from baseline and a 12-week score of <16 points.
Time Frame: 12 weeks after randomization (baseline)
Population: The analysis was limited to participants who completed the 12-week visit within the pre-specified analysis window (10 to 18 weeks, inclusive). Descriptive statistics were performed to compute the number and proportion of participants by treatment group.
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 31
participants | 28 | 25 | 11

4. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria Based on the Mean NPC Break at 12 Weeks by Treatment Group
Description: The number of subjects who are classified as a success based on the mean NPC break at the 12-week visit. Success is based on the mean NPC (near point of convergence) break is defined as having a mean NPC break of <6 cm at 12 weeks and a 12-week to baseline ratio of <0.763 for mean NPC break.
Time Frame: 12 weeks after randomization (baseline)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 31
participants | 33 | 33 | 11

5. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria Based on the Mean PFV Blur at 12 Weeks by Treatment Group
Description: The number of subjects who are classified as a success based on the mean PFV blur at the 12-week visit. Success is based on the mean PFV (positive fusional vergence) blur, defined as having a mean PFV blur of >15 pd at 12 weeks and a 12-week to baseline ratio of >1.419 for mean PFV blur.
Time Frame: 12 weeks after randomization (baseline)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 69
participants | 49 | 35 | 16

6. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria for Both Clinical Measures at 12 Weeks by Treatment Group
Description: The number of subjects classified as a success based on clinical measures of CI (mean NPC break & mean PFV blur) at the 12-week visit. Clinical success is defined according to whether both criteria (below) are met as follows:
  1. Near point of convergence (NPC) break: 12-week/baseline mean NPC break <0.763 and a 12-week mean NPC break <6 cm
  2. Positive fusional vergence (PFV) blur: 12-week/baseline mean PFV blur >1.419 and a 12-week mean PFV blur >15 pd
Time Frame: 12-weeks after randomization (baseline)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 31
participants | 30 | 22 | 9

7. Secondary Outcome: Number of Participants Classified as Having Improved in All 3 Outcomes Measures From Baseline to 12 Weeks by Treatment Group
Description: Improvement in all 3 outcome measures at 12 weeks will be defined as follows:
  1. Convergency Insufficiency Symptom Survey (CISS): Improvement of 9 or more points since baseline
  2. Near point of convergence (NPC) break: 12-week/baseline mean NPC break <0.763
  3. Positive fusional vergence (PFV) blur: 12-week/ baseline mean PFV blur >1.419
  (Note: All 3 criteria must be met in order to be classified as an "improver" at the 12-week primary outcome visit).
Time Frame: 12 weeks after randomization (baseline)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 69 | 69 | 31
participants | 27 | 25 | 10

8. Post Hoc Outcome: Number of Participants Classified as an Overall Success at 12 Weeks in the HB-C Group According to Whether or Not the Computer-based Therapy Program Was Completed at 12 Weeks
Description: This outcome was limited to participants randomly assigned to the HB-C group.
  Completion of the home-based computer therapy program was defined as achieving at least 15 stars on the jump vergence therapy).
  Overall success was defined as meeting the following criteria for all 3 outcome measures at 12 weeks:
  1. Convergence Insufficiency Symptom Survey (CISS): 12-week score of <16 points and at least a 9-point improvement from baseline at 12 weeks
  2. Near point of convergence (NPC) break: 12-week/baseline mean NPC break <0.763 and a 12-week mean NPC break <6 cm
  3. Positive fusional vergence (PFV) blur: 12-week/ baseline mean PFV blur > 1.419 and a 12-week mean PFV blur >15 pd
Time Frame: 12 weeks after randomization (baseline)
Population: The analysis was limited to participants who were randomly assigned to the HB-C group who completed the 12-week visit within the pre-specified analysis window (10 to 18 weeks, inclusive).
Measure: Number; unit: participants
Groups:
- HB-C (Completed Computer-based Therapy Program): Participants in the HB-C treatment group who completed the computer vergence/accommodative therapy (CVAT) program at 12 weeks, defined as achieving at least 15 stars for the jump vergence exercise).
- HB-C (Did Not Complete Computer-based Therapy Program): Participants in the HB-C treatment group who did not complete the computer vergence/accommodative therapy (CVAT) program at 12 weeks, defined as achieving <15 stars for the jump vergence exercise.
Arm/Group | HB-C (Completed Computer-based Therapy Program) | HB-C (Did Not Complete Computer-based Therapy Program)
Number analyzed (Participants) | 22 | 47
participants | 4 | 12
Statistical Analysis 1: Comparison: HB-C (Completed Computer-based Therapy Program); For the HB-C group, the association between completion of the computer vergence/accommodative therapy (CVAT) program (defined as achieving at least 15 stars for the jump vergence exercise) and overall success at 12 weeks was evaluated using Bernard's exact test; Test type: Superiority or Other; p < 0.01, Bernard's exact test; A p-value was not reported in the manuscript results, but has been included here, reported directly from the analysis; Risk Difference (RD) = -7, 95% CI 2-sided [-27 to 17]

9. Secondary Outcome: Number of Participants Classified as an Overall Success Based on the 3 Outcomes Measures From Baseline to 6 Weeks by Treatment Group
Description: To be considered an overall success, each of the following criteria must be met for the 3 outcome measures at 6 weeks:
  1. Convergence Insufficiency Symptom Survey (CISS): 6-week score <16 points and at least 9-point improvement from baseline at 6 weeks
  2. Near point of convergence (NPC) break: 6-week/baseline mean NPC break <0.763 and a mean 6-week NPC break <6 cm
  3. Positive fusional vergence (PFV) blur: 6-week/baseline mean PFV blur >1.419 and a mean 6-week PFV break >15 pd
  (Note: All 3 criteria must be met in order to be classified as an overall success at the 6-week visit).
Time Frame: 6 weeks after randomization (baseline)
Population: The analysis was limited to participants who completed the 6-week visit within the pre-specified analysis window (4 to <10 weeks). Descriptive statistics were performed to compute the number and proportion of participants by treatment group.
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 66 | 71 | 34
participants | 5 | 2 | 1

10. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria Based on CI Signs/Symptoms at 6 Weeks by Treatment Group
Description: The number of subjects classified as a success based on signs/symptoms at the 6-week visit. Success is based on the Convergency Insufficiency Symptom Survey (CISS) defined as improvement of 9 or more points from baseline and a 6-week score of <16 points.
Time Frame: 6 weeks after randomization (baseline)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 66 | 71 | 34
participants | 13 | 8 | 8

11. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria Based on the Mean NPC Break at 6 Weeks by Treatment Group
Description: The number of subjects who are classified as a success based on the mean NPC break at the 6-week visit. Success is based on the mean NPC (near point of convergence) break is defined as having a mean NPC break of <6 cm at 6 weeks and a 6-week to baseline ratio of <0.763 for mean NPC break.
Time Frame: 6 weeks after randomization (baseline)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 66 | 71 | 34
participants | 24 | 20 | 5

12. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria Based on the Mean PFV Blur at 6 Weeks by Treatment Group
Description: The number of subjects who are classified as a success based on the mean PFV blur at the 6-week visit. Success is based on the mean PFV (positive fusional vergence) blur, defined as having a mean PFV blur of >15 pd at 6 weeks and a 6-week to baseline ratio of >1.419 for mean PFV blur.
Time Frame: 6 weeks after randomization (baseline)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 66 | 71 | 34
participants | 38 | 23 | 12

13. Secondary Outcome: Number of Participants Classified as Having Met Success Criteria for Both Clinical Measures at 6 Weeks by Treatment Group
Description: The number of subjects classified as a success based on clinical measures of CI (mean NPC break & mean PFV blur) at the 6-week visit. Clinical success is defined according to whether both criteria (below) are met as follows:
  1. Near point of convergence (NPC) break: 6-week/baseline mean NPC break <0.763 and a 6-week mean NPC break <6 cm
  2. Positive fusional vergence (PFV) blur: 6-week/baseline mean PFV blur >1.419 and a 6-week mean PFV blur >15 pd
Time Frame: 6-weeks after randomization (baseline)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 66 | 71 | 34
participants | 20 | 10 | 3

14. Secondary Outcome: Number of Participants Classified as Having Improved in All 3 Outcomes Measures From Baseline to 6 Weeks by Treatment Group
Description: Improvement in all 3 outcome measures at 6 weeks will be defined as follows:
  1. Convergency Insufficiency Symptom Survey (CISS): Improvement of 9 or more points since baseline
  2. Near point of convergence (NPC) break: 6-week/baseline mean NPC break <0.763
  3. Positive fusional vergence (PFV) blur: 6-week/baseline mean PFV blur >1.419
  (Note: All 3 criteria must be met in order to be classified as an "improver" at the 6-week visit).
Time Frame: 6 weeks after randomization (baseline)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Number analyzed (Participants) | 66 | 71 | 34
participants | 17 | 13 | 3

ADVERSE EVENTS:
Time Frame: 12 week primary outcome.
Arm/Group | Computer-based Therapy (CBT) | Near Target Push-up (NTP) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/85 | 0/44
Other Adverse Events (participants affected / at risk) | 0/75 | 0/85 | 0/44

LIMITATIONS AND CAVEATS:
Differential loss to follow-up (HB-C 8%, HB-PU 19%, and HB-P 30%).

Did not formally assess whether participants remained masked to their treatment group during the study.

Assessment of compliance was not completely objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No